CLINICAL TRIAL: NCT04524819
Title: A Pilot Study to Characterise Saliva and Sputum FTIR Spectral Profiles in Patients with COPD During Exacerbations and When Stable
Acronym: SPIT-D
Status: Terminated | Type: Observational
Why Stopped: Airborne particles during data collection a risk during COVID-19
Sponsor: Portsmouth Hospitals NHS Trust (Other Government)
Responsible Party: Sponsor
Other Study IDs: PHT/2019/46
Record Dates: First submitted 2020-07-10; First posted 2020-08-24 (Actual); Last update posted 2024-11-08 (Actual); Status verified 2024-11

CONDITIONS: Chronic Obstructive Pulmonary Disease
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Sputum and Saliva
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- COPD participants: Saliva and Sputum will be collected from patients when they are unwell with a flare up of the COPS and when they are well

SUMMARY:
This study will characterise saliva and sputum FTIR spectral profiles in patients with COPD, during exacerbations and stable disease.

DETAILED DESCRIPTION:
Chronic Obstructive Pulmonary Disease (COPD) is a common and treatable condition that is characterised by predominately irreversible and progressive airflow limitation. COPD is a leading cause of morbidity and mortality worldwide and its prevalence is predicted to increase substantially in the coming decade1. In the United Kingdom (UK) alone, COPD affects an estimated 3 million people, with 1 million diagnosed and a further 2 million remaining undiagnosed2. Delays in an accurate diagnosis impacts on quality of life and healthcare resource utilisation. COPD is associated with a significant economic and social burden, with a single severe exacerbation requiring admission to hospital costing up to £1600, therefore having a major impact on NHS expenditure. COPD also has a personal burden, causing 24 million lost working days annually, costing the UK economy £3.8 billion3.

Importance is placed on early detection of exacerbations of COPD as delays in starting treatment are associated with increased exacerbation severity, emergency healthcare use, a higher mortality and a more rapid decline in lung function. There is therefore a recognised need for widely accessible, easy-to-use tools to aid in the early detection of COPD exacerbations.

Fourier Transform Infra-Red (FTIR) spectroscopy is an emerging field of medicine which has the potential to become established in the management of lung conditions. Previous studies4,5 have shown that sputum in patients with COPD analysed with infrared (IR) gave reproducible biological IR spectra with distinct signatures in 5 key regions, namely Amide A, two signatures in the Amide I region, Amide II and in glycoproteins. The additional information on the spectral profiles gathered in this study on saliva and sputum from patients with COPD, during both stable disease and exacerbations will help establish FTIR use in the management of these lung conditions.

This study will provide essential information in the development process of a hand held FTIR spectroscope. Phase 1 will establish the infrared spectrum required for the analysis of saliva and sputum, which will inform the design of the daisy chain device (a pre-prototype device) used in phase 2. Phase 2 will test this infrared spectrum in the pre-prototype daisy chain device with further saliva and sputum samples, before this spectrum is incorporated into the eventual hand-held FTIR spectroscope.

ELIGIBILITY:
Inclusion Criteria:

* Participants with a confirmed diagnosis of an exacerbation of COPD (aged ≥40 years), n=40 (20 participants recruited in phase 1 and 20 participants recruited in phase 2) who are able to spontaneously expectorates sputum during exacerbations and on at least 3 out of 7 days when well.
* Able to provide written informed consent

Exclusion Criteria:

* Participants with other significant respiratory disease that, in the opinion of the clinical investigator, is the major cause of their respiratory symptoms (e.g. pulmonary tuberculosis, allergic bronchopulmonary aspergillosis, pulmonary fibrosis).
* Participants with COPD whose deterioration in respiratory symptoms is not thought to be due to an exacerbation of their COPD (e.g. pneumonia*, pneumothorax, pulmonary embolus).

  * A member of the research study medical team will review the participant's chest X-Ray (CXR) to exclude any pneumonia, defined by consolidation on CXR before they are recruited onto the study if a CXR has been taken. In participants who have not had a CXR, exclusion of pneumonia will be based on clinical assessment.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants with COPD
Sampling Method: Non-Probability Sample
Enrollment: 27 (Actual)
Dates: Start 2019-09-18 (Actual); Primary Completion 2023-10-31 (Actual); Study Completion 2023-10-31 (Actual)

PRIMARY OUTCOMES:
Disease severity | within a 24 month period
  measured using the GOLD refined ABCD Assessment Tool
Disease Control | a change between the exacerbation visit and stable visit through study completion, an average of 2 years
  measured using the COPD Assessment Tool
FEV1 forced expiratory volume-one second | a change between the exacerbation visit and stable visit through study completion, an average of 2 years
  Assessment of lung function using spirometry to measure lung airflow
FVC forced vital capacity | a change between the exacerbation visit and stable visit through study completion, an average of 2 years
  Assessment of lung function using spirometry to measure lung airflow
FEV1/FVC ratio | a change between the exacerbation visit and stable visit through study completion, an average of 2 years
  Assessment of lung function using spirometry to measure lung airflow
Sputum Culture | immediately during analysis
  FTIR wavelength

CONTACTS AND LOCATIONS:
Locations (1):
- Portsmouth Hospitals NHS Trust, Queen Alexandra Hospital, Portsmouth, Hampshire, United Kingdom

IPD SHARING:
Plan to Share IPD: No